CLINICAL TRIAL: NCT03614468
Title: New Infant Formula Supports Adequate Growth and Safety Study in Healthy Infants
Brief Title: New Infant Formula Supports Adequate Growth in Healthy Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Worthy Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 79105203
Record Dates: First submitted 2018-07-17; First posted 2018-08-03 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Infant Development
Keywords: Infant Formula

STUDY DESIGN:
Intervention Model Description: Formula feed infants will be randomized to receive either a new infant formula formulated for healthy term infants (Formula A) or a commercially available infant formula for healthy term infants (Formula B). Infants will consume the formula for a total of 52-weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a randomized, controlled, double-blind, study of healthy term formula fed (FF) infants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Formula A (Experimental): An experimental Infant Formula, Milk-Based Powder with Iron, for healthy term infants 0 to 12 months of age.
  Interventions: Other: Formula A
- Formula B (Active Comparator): A Commercially available Infant Formula, for healthy term infants 0 to 12 months of age (Enfamil TM, Milk-Based Powder with Iron)
  Interventions: Other: Formula B

INTERVENTIONS:
Other: Formula A — Formula A is to be feed as the sole source of nutrition for 52 weeks to healthy term infants.
  Arms: Formula A
Other: Formula B — Formula B is to be feed as the sole source of nutrition for 52 weeks to healthy term infants.
  Arms: Formula B

SUMMARY:
The objective of the present study is to evaluate the growth, safety, and tolerance in healthy, term infants consuming a new to market infant formula (Formula A) and a commercially available infant formula (Formula B) with daily weight gain as the primary outcome. As secondary outcomes, the study will evaluate other growth parameters, tolerance, and safety.

DETAILED DESCRIPTION:
This is a controlled randomized parallel assignment, masked (Participant, Care Provider, Investigator, Outcomes Assessor) study. Healthy infants will be assigned an Investigational (Formula A) experimental new milk based infant formula, or an active comparator Control (Formula B) Enfamil (trademark brand name) marketed milk based infant formula. The period for the study is 365 days (52 weeks) using repeated-measures mixed model (RMMM). Anthropometry, formula intake, tolerance, and stool characteristics will be assessed. Medically confirmed adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Infants will be eligible to participate if they meet all of the following conditions. At birth the infant must be:

Only infants whose parent(s) or legal guardian(s) have decided to feed infant formula as the sole source of nutrition, will be approached for potential study enrollment

1. Healthy, term (early term/no less than 37 weeks, 0 days through late term/no greater than 41 weeks, 6 days), singleton infant
2. Have a birth weight of ≥ 2500 grams

At the time of the baseline/enrollment visit, infants must be:

1. Designated as healthy by a physician
2. ≤21 days post-natal age (Date of Birth = Day 0)
3. Weight for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
4. Length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
5. Head circumference for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
6. Weight for length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
7. Exclusively consuming and tolerating a cow's milk infant formula at time of enrollment
8. Have parent(s) or legal guardian(s) who agree to feed the study formula to the study subject as his/her sole source of nutrition for the duration of the study
9. Have parent(s) or legal guardian(s) who have read and voluntarily signed an Informed Consent form approved by the Institutional Review Board prior to any participation in the study.

Exclusion Criteria:

Infants will be ineligible if they have any of the following conditions that are judged by a physician to interfere with the infant's normal growth, development, and/or tolerance to an infant formula:

1. Infants showing evidence of anatomic and physiologic defects of the respiratory tract, or other congenital defects (as determined by the clinician)
2. Evidence of chronic hepatic, gastrointestinal, renal, cardiac, pulmonary, or neurological diseases
3. Having a maternal history with known adverse effects on the fetus and/or the newborn infant, such as diabetes (gestational diabetes is acceptable if infant's birth weight is < 4300 g), active tuberculosis, perinatal infection,
4. Having a family history of cow's milk protein intolerance/allergy
5. Are an infant from a multiple birth (twin, triplet, etc.)
6. Mothers who smoked cigarettes
7. Mothers who used illicit drugs during pregnancy.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-05-08 (Estimated); Primary Completion 2020-05-08 (Estimated); Study Completion 2020-05-25 (Estimated)

PRIMARY OUTCOMES:
Weight gain change measured at set intervals for first 365 days | 1-21 days, 42 days, 84 days, 126 days, 180 days, 270 days, 365 days
  The infants will be weighed naked while lying quietly on a calibrated electronic scale accurate to 10 grams.

SECONDARY OUTCOMES:
Safety and Tolerability evaluated and recorded by parents in daily journal on stool observations at start through 365 days using VAS (Visual Analogue Scale) | Daily through 365 days
  1. Daily stool frequency
  2. Stool consistency (on a five-point scale: 1 = watery, 2 = soft/pudding like, 3 = soft formed, 4 = dry formed, 5 = dry/hard pellets)
  3. Constipation (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  4. Diarrhea (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  5. Colic (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  6. Vomiting (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  7. Regurgitation (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  8. Flatulence (0 = absent, 1 = mild, 2 = moderate, 3 = severe)
  9. Nappy rash (0 = absent, 1 = mild, 2 = moderate, 3 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Worthy, Study Director — Chairman, Worthy Health

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be publicly available containing the abstract, background, materials and methods, study design, procedures, study formulas, measurements, statistics, results, adverse events, discussion, acknowledgements, and references.

REFERENCES:
- [Result] Field CJ. The immunological components of human milk and their effect on immune development in infants. J Nutr. 2005 Jan;135(1):1-4. doi: 10.1093/jn/135.1.1. PMID 15623823
- [Result] Garcia C, Duan RD, Brevaut-Malaty V, Gire C, Millet V, Simeoni U, Bernard M, Armand M. Bioactive compounds in human milk and intestinal health and maturity in preterm newborn: an overview. Cell Mol Biol (Noisy-le-grand). 2013 Dec 30;59(1):108-31. PMID 25326648
- [Result] Jost T, Lacroix C, Braegger C, Chassard C. Impact of human milk bacteria and oligosaccharides on neonatal gut microbiota establishment and gut health. Nutr Rev. 2015 Jul;73(7):426-37. doi: 10.1093/nutrit/nuu016. Epub 2015 Apr 15. PMID 26081453
- [Result] Koletzko B, Baker S, Cleghorn G, Neto UF, Gopalan S, Hernell O, Hock QS, Jirapinyo P, Lonnerdal B, Pencharz P, Pzyrembel H, Ramirez-Mayans J, Shamir R, Turck D, Yamashiro Y, Zong-Yi D. Global standard for the composition of infant formula: recommendations of an ESPGHAN coordinated international expert group. J Pediatr Gastroenterol Nutr. 2005 Nov;41(5):584-99. doi: 10.1097/01.mpg.0000187817.38836.42. PMID 16254515
- [Result] Verwimp JJ, Bindels JG, Barents M, Heymans HS. Symptomatology and growth in infants with cow's milk protein intolerance using two different whey-protein hydrolysate based formulas in a Primary Health Care setting. Eur J Clin Nutr. 1995 Sep;49 Suppl 1:S39-48. PMID 8647062
- [Result] Szajewska H, Chmielewska A. Growth of infants fed formula supplemented with Bifidobacterium lactis Bb12 or Lactobacillus GG: a systematic review of randomized controlled trials. BMC Pediatr. 2013 Nov 12;13:185. doi: 10.1186/1471-2431-13-185. PMID 24215626
- [Result] Saha KK, Frongillo EA, Alam DS, Arifeen SE, Persson LA, Rasmussen KM. Use of the new World Health Organization child growth standards to describe longitudinal growth of breastfed rural Bangladeshi infants and young children. Food Nutr Bull. 2009 Jun;30(2):137-44. doi: 10.1177/156482650903000205. PMID 19689092